CLINICAL TRIAL: NCT04502914
Title: The Study on Bacterial Load Following Open-to-air Management in Burn Patients.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of subjects enrolled
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB #: L20-067
Record Dates: First submitted 2020-07-29; First posted 2020-08-06 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Burns; Infection Wound; Bacterial Infections
MeSH Terms: conditions — Burns; Wound Infection; Bacterial Infections

STUDY DESIGN:
Intervention Model Description: The experimental group will consist of wounds treated with the open-to-air strategy. The control group will consist of wounds treated with traditional closed-wound management with dressings soaked in topical antimicrobial solutions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The experimental group (Experimental): The experimental group will consist of wounds treated with the open-to-air strategy.
  Interventions: Procedure: Open-to-air strategy
- The control group (Other): The control group will consist of wounds treated with traditional closed-wound management with dressings soaked in topical antimicrobial solutions.
  Interventions: Procedure: Traditional closed-wound management

INTERVENTIONS:
Procedure: Open-to-air strategy — In open-to-air management, the wound will be washed with a chlorhexidine solution and leave the wound open, or portion of the wound assigned to OTA, to the environment. An electric heat lamp (model no. 53103, 250W, Brandt Industries LLC, Bronx, NY) will be placed at as close to 1 yard (0.91 m) as possible from the wound after daily wound care for 24 hours (+/- 6 hours) to promote drying. However, to prevent excessive drying an hourly spritz of topical solution, e.g., DuoDERM® Hydroactive® gel (ConvaTec Oklahoma City, OK) will be used at the bedside.
  Arms: The experimental group
Procedure: Traditional closed-wound management — In traditional closed-wound management, once a day the wound will be washed with a chlorhexidine solution and closed with a non-adherent dressing such as ADAPTIC® (Acelity, San Antonio, TX) soaked in topical antimicrobial solutions, ointments, and creams designed to promote wound healing.
  Arms: The control group

SUMMARY:
Burns are one of the common forms of trauma and are a cause of unintentional death and injury. Management of burns becomes complex due to multiple associated complications, for instance, secondary infection of burn wounds is the most common complication associated with burn injuries. Treatment of bacterial infections with antibiotics is becoming more challenging due to the development of multidrug-resistance. Hence, there is a critical need to investigate and establish non-antibiotic approaches to prevent colonization, control growth, and eliminate bacteria from burn wounds. Recent studies have explored the beneficial effects of open-to-air strategies on wound healing. Based on the evidence, the investigators hypothesize that bacterial load in burn wounds will be lowered when treated with an open-to-air strategy compared to the traditional closed wound approach.

DETAILED DESCRIPTION:
Burns are one of the common forms of trauma and are a cause of unintentional death and injury in the world as well as in the United States (US). Management of burns becomes complex due to multiple associated complications, which result in short-term and long-term disability. Secondary infection of burn wounds is the most common complication associated with burn injuries. Approximately 10,000 people die in the US due to burn-related infections. For instance, gram-negative Pseudomonas aeruginosa is an opportunistic organism commonly found in burn wounds. Bacterial infections cause prolonged hospital stay, increase morbidity, and mortality of burn patients. Treatment of bacterial infections with antibiotics is becoming more challenging due to the development of multidrug-resistance. Hence, current antibiotic regimens and wound care are not always successful in eliminating bacterial infections. As such, there is a critical need to investigate and establish non-antibiotic approaches to prevent colonization, control growth, and eliminate bacteria from burn wounds.

Recent studies have explored the beneficial effects of open-to-air strategies on wound healing, especially in the presence of necrotizing infections. In an open-to air strategy, the wound is left open to the external environment with a heat lamp placed at 6 feet to promote drying. However, the spritz of a topical solution will be applied to avoid excessive drying. Based on current evidence, the investigators hypothesize that bacterial load in burn wounds will be lowered when treated with an open-to-air strategy compared to the traditional closed wound approach.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 89
2. Burn patients with TBSA≥ 20%
3. Any suspicion of skin colonization or infection based on a positive result of microbiologic testing. Testing would only be performed if the attending surgeon treating the patient had a clinical suspicion of wound infection.

Exclusion Criteria:

1. Children

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-06-09 (Actual); Study Completion 2021-06-09 (Actual)

PRIMARY OUTCOMES:
The bacterial load at baseline for each treatment | At baseline
  Scrapings of the superficial wound exudate and debris will be obtained at baseline (i.e., the 0-time point before implementing any the tested wound care management option) from both wound sites of each patient.
  The colony-forming units (CFUs) will be enumerated and CFUs/g will be calculated for treatment and control.
The bacterial load on day 1 for each treatment | On day 1
  Scrapings of the superficial wound exudate and debris will be obtained on day 1 (about 24 hours after obtaining samples for baseline measurement) from both wound sites of each patient.
  The colony-forming units (CFUs) will be enumerated and CFUs/g will be calculated for treatment and control.
The bacterial load on day 2 for each treatment | On day 2
  Scrapings of the superficial wound exudate and debris will be obtained on day 2 (about 48 hours after obtaining samples for baseline measurement) from both wound sites of each patient.
  The colony-forming units (CFUs) will be enumerated and CFUs/g will be calculated for treatment and control.
Difference in change in bacterial load for day 1 | Change in bacterial load from baseline and day 1
  Change in bacterial load from baseline and day 1 and compared between treatment and control groups.
Difference in change in bacterial load for day 2 | Change in bacterial load from baseline and day 2
  Change in bacterial load from baseline and day 2 and compared between treatment and control groups.

SECONDARY OUTCOMES:
Prevalence of bacterial species at baseline for each treatment | At baseline
  Scrapings of the superficial wound exudate and debris will be obtained at baseline from both wound sites of each patient.
  Debridement samples will be homogenized and serially diluted.The dilutions will be spot plated on selective agar.
Prevalence of bacterial species on day 1 for each treatment | On day 1
  Scrapings of the superficial wound exudate and debris will be obtained at baseline on day 1 from both wound sites of each patient.
  Debridement samples will be homogenized and serially diluted.The dilutions will be spot plated on selective agar.
Prevalence of bacterial species on day 1 for each treatment | On day 2
  Scrapings of the superficial wound exudate and debris will be obtained on day 2 from both wound sites of each patient.
  Debridement samples will be homogenized and serially diluted.The dilutions will be spot plated on selective agar.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Tech University Health Sciences Center, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yang D, Davies A, Burge B, Watkins P, Dissanaike S. Open-to-Air Is a Viable Option for Initial Wound Care in Necrotizing Soft Tissue Infection that Allows Early Detection of Recurrence without Need for Painful Dressing Changes or Return to Operating Room. Surg Infect (Larchmt). 2018 Jan;19(1):65-70. doi: 10.1089/sur.2017.080. Epub 2017 Dec 6. PMID 29211657
- [Result] Dai T, Gupta A, Huang YY, Yin R, Murray CK, Vrahas MS, Sherwood ME, Tegos GP, Hamblin MR. Blue light rescues mice from potentially fatal Pseudomonas aeruginosa burn infection: efficacy, safety, and mechanism of action. Antimicrob Agents Chemother. 2013 Mar;57(3):1238-45. doi: 10.1128/AAC.01652-12. Epub 2012 Dec 21. PMID 23262998